CLINICAL TRIAL: NCT06800144
Title: Effect of Telerehabilitation-Based Heart Rate-Synchronized Motor Imagery Music Therapy on Pain, Autonomic Function and Psychosocial Parameters in People With Multiple Sclerosis
Brief Title: Effect of Music Therapy on Pain in People With Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Hilal Karakas, Research Assistant, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MusicTherapy
Record Dates: First submitted 2025-01-20; First posted 2025-01-29 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis, MS
Keywords: Music Therapy in Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Heart rate synchronized motor imagery music therapy (Experimental): Participants included in this group will imagine the movements presented to them with a metronome sound in a rhythm synchronized with their heart rate.
  Interventions: Behavioral: Heart rate synchronized motor imagery music therapy
- Heart rate synchronized music therapy (Active Comparator): Participants included in this group will listen to soothing/relaxing music without lyrics in a rhythm synchronized with their heart rate.
  Interventions: Behavioral: Heart rate synchronized music therapy
- Control group (No Intervention): Participants included in this group will continue their routine treatment and will only be evaluated three times: at the beginning, after 8 weeks and after 12 weeks.

INTERVENTIONS:
Behavioral: Heart rate synchronized motor imagery music therapy — Participants included in this group will listen a metronome sound in a rhythm synchronized with their heart rate.
  Arms: Heart rate synchronized motor imagery music therapy
Behavioral: Heart rate synchronized music therapy — Participants included in this group will listen to soothing/relaxing music without lyrics in a rhythm synchronized with their heart rate.
  Arms: Heart rate synchronized music therapy

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory, demyelinating and progressive neurological disease of the central nervous system, often seen between the ages of 20-30. Pain is a very common symptom in people with MS, with a prevalence of 63%. Pain in MS is a symptom that negatively affects individuals' fatigue, anxiety and depression levels, quality of life and sleep quality. In addition, chronic pain affects individuals' autonomic and cognitive functions. Music therapy is defined as the systematic use of music in a therapeutic relationship that aims to improve, maintain and develop emotional, physical and mental health. Music therapy protocols synchronized with heart rate can be effective on chronic pain through the regulation of the autonomic nervous system and activation of the parasympathetic nervous system. Studies indicate that music therapy, regardless of the population applied, is effective in the management of symptoms such as pain, depression and anxiety. Motor imagery training is a method that regulates cerebral cortex activity by exposing the brain to visual information and imagination, reduces abnormal cortical activation, and thus restores the brain's ability to change. Research indicates that the most effective motor imagery training in reducing pain is motor imagery training presented in a protocol graded from simple to complex motor tasks.

The grading principle applied in motor imagery training in the form of imagining movements from simple to complex and music therapy training presented in a rhythm matched with heart rate rhythm are effective approaches on chronic pain. It is thought that the treatment protocol in which these two methods are combined and their therapeutic effects are combined in MS rehabilitation may be more effective on pain and related factors in MS. The aim of the study is to show the effects of telerehabilitation-based heart rate-synchronized music therapy protocols on pain, heart rate, fatigue, anxiety, depression, quality of life, sleep quality, and information processing speed compared to MS individuals who continue their routine treatments.

45 MS people with chronic pain will be included in the planned randomized controlled trial. The included participants will be randomized into 3 groups with 15 participants in each group. The evaluations will be performed three times before treatment, at 8th (post-treatment evaluation) and 12th weeks (follow-up evaluation). The participants' general pain intensity in the last 2 and 7 days, the presence of neuropathic pain, fatigue level, anxiety and depression levels, sleep quality, health-related quality of life and information processing speed will be evaluated. In addition, heart rate variability will be evaluated in order to evaluate the participants' autonomic functions. Telerehabilitation-based music therapy application will be given to the participants 2 days a week for 8 weeks using a videoconferencing platform under the guidance of a physiotherapist. The heart rates of the participants will be monitored throughout the session. The participants included in the first group will visualize the movements presented with the metronome sound in a rhythm matched to their heart rates, while the participants included in the second group will listen to relaxing/relaxing music without lyrics in a rhythm matched to their heart rates. When synchronization is achieved between the music rhythm and the heart rate in both groups, the music rhythm will be reduced. Participants included in the 3rd group will continue their routine treatment and will be evaluated only three times: at the beginning, after the 8th week and after the 12th week. The results obtained from this study will examine the effects of heart rate synchronized music therapy protocols on pain, autonomic function and psychosocial parameters in individuals with chronic pain and MS.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65.
* Having a definite MS diagnosis according to the 2017 McDonald criteria.
* Having a pain level of at least 3 and above on the numerical pain scale for at least 3 months.
* Not having had an attack in the last 3 months.
* Having a tablet or computer with an active internet connection that is suitable for videoconferencing.
* Having a smartphone to which the heart rate monitor can be connected with the Bluetooth feature so that the heart rate synchronized music therapy training can be given.
* Having sufficient smartphone/tablet or computer knowledge to participate in the study or having a relative who can help in this regard.
* No change in the medications used for pain in the last 2 months.
* Not receiving any additional treatment other than routine treatments.
* Being able to read and understand Turkish.

Exclusion Criteria:

* Having a serious musculoskeletal, cardiovascular, pulmonary, metabolic or other disease that would prevent participation in the study.
* Having a condition other than MS that can cause pain, such as cancer, diabetes, significant osteoarthritis or rheumatoid arthritis, based on laboratory or imaging findings
* Having a psychiatric disease (such as active psychotic disorders, severe depression, anxiety disorders) that would prevent participation in the study and having a serious cognitive disorder determined by a physician that would prevent testing
* Having a serious vision or hearing problem.
* Being pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, week 8 and week 12
  The general pain intensity felt by people with MS participating in the study in the last 2 and 7 days will be assessed using the Visual Analogue Pain Scale. The scale ranges from 0 mm to 100 mm, with higher values indicating greater pain intensity.

SECONDARY OUTCOMES:
PainDETECT | Baseline, week 8 and week 12
  'PainDETECT' will be used to assess neuropathic pain in people with MS participating in the study.
Nordic Musculoskeletal Questionnaire | Baseline, week 8 and week 12
  The 'Nordic Musculoskeletal Questionnaire' will be used to assess the pain of MS patients participating in the study according to their body regions.
Central Sensitization Questionnaire- Short Form | Baseline, week 8 and week 12
  The Central Sensitization Questionnaire-Short Form is a participant-reported measurement tool designed to assess the presence of central sensitization and its associated symptoms.
Modified Fatigue Impact Scale | Baseline, week 8 and week 12
  The 'Modified Fatigue Impact Scale', which is frequently used in clinical and experimental studies, will be used to determine the fatigue level of people with MS participating in the study. The scale ranges from 0 to 84, with higher values representing increased levels of fatigue.
Hospital Anxiety and Depression Scale | Baseline, week 8 and week 12
  The 'Hospital Anxiety and Depression Scale' will be used to evaluate the anxiety and depression levels of people with MS participating in the study. The questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Preference Based MS Index | Baseline, week 8 and week 12
  The Preference-Based MS Index will be used to assess patient-reported health-related quality of life.
Pittsburgh Sleep Quality Index | Baseline, week 8 and week 12
  The subjective sleep quality of individuals with MS participating in the study will be evaluated using the 'Pittsburg Sleep Quality Index (PSQI)'.
Heart Rate Variability | Baseline, week 8 and week 12
  Heart rate variability is an important parameter of cardiac autonomic modulation and provides information about the autonomic nervous system functions of individuals.
Paced Auditory Serial Addition Test | Baseline, week 8 and week 12
  Paced Auditory Serial Addition Test (PASAT) will be used to assessment the cognitive functions of the participants included in the study.

IPD SHARING:
Plan to Share IPD: No